CLINICAL TRIAL: NCT02972684
Title: Cost-Utility Analysis of Management of Peri Operative Haemorrhage Following Cardiac Surgery Using Conventional Blood Coagulation Tests or Thrombo-elastographic Point of Care Test - IMOTEC
Brief Title: Cost-Utility Analysis of Management of Peri Operative Haemorrhage Following Cardiac Surgery With Cardiopulmonary Bypass
Acronym: IMOTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC16_0009
Record Dates: First submitted 2016-11-02; First posted 2016-11-23 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: C.Surgical Procedure; Cardiac; Blood Transfusion; Blood Coagulation Disorders; Bypass, Cardiopulmonary; Hemostatic
Keywords: Cardiopulmonary Bypass; Hemorrhage; blood transfusion; Point-of-care test; health economics
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional coagulation management (No Intervention): management of perioperative haemorrhage following cardiac surgery using conventional blood coagulation tests.
- Thrombo-elastometry POC testing (Experimental): management of perioperative haemorrhage following cardiac surgery using the thrombo-elastometry point of care test.
  Interventions: Device: Thrombo-elastometry POC testing

INTERVENTIONS:
Device: Thrombo-elastometry POC testing — Use of thrombo-elastometry point of care test and algorithm guided predetermined intervention during peri operative haemorrhage
  Arms: Thrombo-elastometry POC testing

SUMMARY:
Peri operative haemorrhage following cardio Pulmonary Bypass may occur in 5 to 10% of cardiac surgical interventions.

Treatment of such complication often necessitates various combinations therapeutic intervention including allogenic blood products administration, drug use and/or surgical intervention. All are expensive treatment and decision making is guided by patient clinical status and biological tests of the haemostatic function.

A key point is the time frame of the clinical process. Therapeutic choices have to be done as fast as possible to minimize bleeding consequences on patient haemodynamic and physiological status. Conventional coagulation test results availability time usually exceed 45' after blood drawing. In such situation, the results may not reflect precisely the coagulation system current state. This downside is often counterbalanced by clinicians empirical choices preceding lab test results knowledge that may conduct to inappropriate treatment, blood product overuse and undue expense.

Viscoelastic point of care test may compensate for the limitations of conventional coagulation tests. In perioperative haemorrhage, faster and more precise information about haemostatic function may help for more accurate therapeutic choices.

The IMOTEC study aims to compare haemorrhage management following cardiac surgery using conventional blood coagulation tests or thrombo-elastogaphic point of care test.

Primary endpoint is a cost utility analysis of the technology and secondary endpoints include blood component transfusion, postoperative bleeding , thoracic re-intervention, postoperative infection (any cause), organ failure, in hospital length of stay and death.

DETAILED DESCRIPTION:
The research is a real life, prospective, single blinded stepped wedge randomized study.

Inclusion after informed consent of adult patient having cardio-vascular surgical procedure using cardiopulmonary bypass and meeting inclusion criterion "bleeding".

After meeting inclusion criterion patients are managed either using conventional blood coagulation tests or using thrombo-elastometry POC test and predefined therapeutic interventions described in a specific algorithm.

Other elements of patient clinical management follow usual center standard care .

Follow up of EQ-5D and clinical evaluations are performed at one , 6 and 12 months after inclusion.

ELIGIBILITY:
Pre-Inclusion Criteria:

* Adult patients over 18 years old scheduled for elective or urgent cardiac surgery using cardiopulmonary bypass .
* Patient informed written consent (non-opposition to data use) or person of trust or family member information .

Inclusion Criteria:

Blood Coagulation test sampling indication for intra or post-operative bleeding defined as follow:

1. intra-operative post CPB bleeding; evaluation more than 10min after heparin reversal by protamin.

   * Clinically significant bleeding judged on surgeon and anesthesiologist consensual point of view
   * Sternal closure delay
   * Chest tube bleeding exceeding 50ml in 10min or more than 1ml/kg in 30min (2ml/kg/h)
2. Postoperative period , evaluation in post operative care environment after 30min stabilization period

   * Chest tube bleeding exceeding 50ml in 10min or more than 1ml/kg in 30min (2ml/kg/h)
   * Patient requiring surgical re-exploration for diagnosed or suspected pericardial effusion or surgical site bleeding requiring surgical hemostatic intervention

Exclusion Criteria:

* Known congenital bleeding disorder
* Redo surgery for patient previously included in the study
* Implantation of Cardiac support device, Extra Corporeal Membrane Oxygenation (ECMO) Extra Corporeal Life support (ECLS), uni or bi-ventricular artificial hearts.
* Indication for post-CPB ECMO or ECLS
* blood transfusion refusal
* pregnant women
* patients under 18 years old
* Adult patient under guardianship, trusteeship or safeguard justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1098 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Cost-utility ratio | one year
  incremental cost per incremental life year and incremental costs per incremental QALY

SECONDARY OUTCOMES:
incremental cost effectiveness ratio | one year
  incremental cost effectiveness ratio : difference in costs divided by the difference in mortality and serious adverse events
Complication rates | one year
  Parameters followed during hospitalization are: volume of postoperative bleeding, allogeneic blood product transfusion, blood cell count, postoperative complications: surgical reexploration, acute kidney injury, need for renal replacement therapy, organ failure, acquired infections, mechanical ventilation duration, intensive care, and in hospital length of stay, death.
Complication rates | one year
  The major complications that can occur within 12 months are: death, cardio-thoracic surgical intervention, acute kidney injury, need for renal replacement therapy, any serious illness diagnosis.
Evaluation survey | Day 1
  Evaluation survey regarding the context and the parameters that impacted the physician's decision, which will be used a sub-group of 100 patients.
The location of the Thrombo-elastometry POC testing | three years
  The location of the Thrombo-elastometry POC testing (operative room or laboratory)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Rozec, PUPH, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - Angers University Hospital, Angers
  - Bordeaux University hospital, Bordeaux
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Dijon University Hospital, Dijon
  - Lille University hospital, Lille
  - Marseille AP-HM La Timone, Marseille
  - Nancy University Hospital, Nancy
  - APHP, La Pitié Salpétrière, Paris
  - HEGP, Hôpital Européen Georges Pompidou, Paris
  - Rouen University Hospital, Rouen
  - Saint-Etienne University Hospital, Saint-Etienne
  - Strasbourg Universtiy Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigal JC, Boissier E, Lakhal K, Riche VP, Durand-Zaleski I, Rozec B. Cost-effectiveness of point-of-care viscoelastic haemostatic assays in the management of bleeding during cardiac surgery: protocol for a prospective multicentre pragmatic study with stepped-wedge cluster randomised controlled design and 1-year follow-up (the IMOTEC study). BMJ Open. 2019 Nov 5;9(11):e029751. doi: 10.1136/bmjopen-2019-029751. PMID 31694845
- [Derived] Vourc'h M, Boissier E, Lakhal K, Grosjean S, Labaste F, Robin E, Bougle A, Mattei M, Morel J, Wurtz V, Mertes PM, Zlotnik D, Lagier D, Beurton A, Rineau E, Fischer MO, May MA, Medard A, Guimbretiere G, Durand-Zaleski I, Pere M, Rozec B, Rigal JC. Cost-utility of point-of-care viscoelastic hemostatic assays in the management of bleeding during cardiac surgery: a single-blinded prospective multicenter stepped wedge cluster randomized trial in French context. Anaesth Crit Care Pain Med. 2025 Nov 20:101704. doi: 10.1016/j.accpm.2025.101704. Online ahead of print. PMID 41274376